CLINICAL TRIAL: NCT05539625
Title: Mitochondrial Antioxidant Therapy to Resolve Inflammation in Ulcerative Colitis (Mini-MARVEL): A Phase 2b Feasibility Randomised Placebo Controlled Trial of Oral MitoQ in Mild-tomoderately Active Paediatric UC
Brief Title: Mini-MARVEL - Mitochondrial Antioxidant Therapy in Ulcerative Colitis
Acronym: Mini-MARVEL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to secure IMP supply.
Sponsor: University of Edinburgh (Other)
Collaborators: The Jon Moulton Charity Trust (Unknown); MitoQ (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AC21067
Record Dates: First submitted 2022-08-04; First posted 2022-09-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ (Active Comparator): Once daily dosing of two capsules for 40mg/d (or one capsule for 20mg/d if weight <30kgs)
  Interventions: Dietary Supplement: MitoQ
- Placebo (Placebo Comparator): Participants will take an oral matched placebo daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MitoQ — MitoQ in inflammation: In the experimental setting, MitoQ has been extensively studied with clear mode of action on inflammatory mechanisms relevant to IBD:
  MitoQ can limit the damage to mitochondria caused by mitochondrial ROS and thereby reducing the leak and oxidisation of mtDNA that are critical to its pro-inflammatory actions within the cell.
  MitoQ reduces the inflammatory potential of mitochondrial DNA which have escaped or released from dying inflammatory cells.
  MitoQ can influence how the immune cells generate their energy, diverting it away from a more inflammatory type of metabolism (glycolysis) MitoQ can induce autophagy, a cellular recycling mechanism that removes damaged mitochondria. Defective autophagy is heavily implicated in the pathogenesis of IBD.
  Hence collectively, MitoQ acts upstream of several pro-inflammatory mechanisms with the net effect to promote resolution of inflammation and mucosal healing.
  Arms: MitoQ
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Mini-MARVEL study, children and young people with an active flare of UC requiring either the start of or an increase in existing mesalazine therapy will be given either MitoQ or placebo as a daily capsule for 24 weeks in the Mini-MARVEL M arm of the study. Those children and young people with an active flare of UC requiring the start of an oral steroid course will be given either MitoQ or placebo as a daily capsule for 24 weeks in the Mini- MARVEL S arm of the study, Further, newly diagnosed children and young people with UC can have either MitoQ or placebo as a daily capsule for 24 weeks with their newly started mesalazine therapy in the Mini-MARVEL M arm of the study, or with their newly started oral steroid course in the Mini-MARVEL S arm of the study. This trial will look at how feasible a multi-centre stratified RCT of this add-on (adjunct) therapy in paediatric UC is in the UK. An assessment after 6, 12 and 24 weeks will be carried out to find out if MitoQ will result in higher rates of improvement in the participants' symptoms, quality of life and gut lining inflammation. Furthermore, the trial will investigate if their UC will be better controlled and that they are less likely to need further steroids or more potent forms of drugs.

MitoQ has been shown to be safe in 2 large human clinical studies in Parkinson's disease and Hepatitis C, but the Mini-MARVEL study, starting alongside the adult MARVEL study, will be the first study in UC in children and young people. At low doses, MitoQ is used as a nutritional supplement that has an anti-oxidant effect. Currently, many drug treatments in UC are very strong, expensive and aimed at suppressing the immune system. Steroid courses are often needed but these have lots of adverse events in children and young people and are strongly disliked by many. If the Mini- MARVEL study provides supportive data on feasibility, including where we have to concentrate our efforts to include enough children and young people through to study end, we could design a full-scale trial to see if MitoQ can be a safe and cost-effective new treatment that works at blocking the specific inflammatory signal found in the gut lining of children and young people with UC.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to17 years in a PIBD service
* Able and willing to give informed consent if aged 16-17 years of age; parents or guardian able and willing to give informed consent if a child of age 15 years and under
* Confirmed UC as documented in the medical notes
* Mild-moderate severity (PUCAI score 10-55)
* (i) If Incident (newly diagnosed) case (biopsy confirmation of suspected UC at endoscopy) or within 2 weeks of diagnosis - no anti-inflammatory medication or if started on 5-ASA on day of endoscopy for presumed UC (ii) If Prevalent case - No medication or stable dose of existing medicine (oral/topical 5-ASA for >2 weeks at screening; thiopurine for >4 weeks at screening)

Exclusion Criteria:

* Inability to swallow capsules
* Young person (16-17 years of age) with inability to provide consent due to a lack of capacity
* Crohn's disease (CD) or IBD unclassified (IBDU) as documented in the medical notes
* Evidence of acute severe UC (ASUC) - ASUC is a medical emergency in children and young people with UC who are clinically unwell with marked diarrhoea, haematochezia and abdominal pain, and by definition have a paediatric UC activity index (PUCAI) score of at least 65 points
* Physician judgement that the subject is likely to require hospitalisation for medical care or surgical intervention of any kind for UC (e.g. colectomy) within 12 weeks of baseline
* Evidence of current (or previous in last 12 months) toxic megacolon (using defined paediatric criteria - radiographic evidence of transverse colon diameter ≥56 mm (or >40mm in those <10 years) PLUS evidence of systemic toxicity (such as: fever >38 degrees Celsius, tachycardia (heart rate >2 SD above mean for age), dehydration, electrolyte disturbance (sodium, potassium or chloride), altered level of consciousness, coma, hypotension or shock) or bowel perforation
* Infective colitis in UC (C&S, C. difficile toxin positive or virology at screening)
* Proctitis (inflammation confined to the rectum, with no proximal extension to the sigmoid) for incident cases after colonoscopy or prevalent cases at most recent colonoscopy
* UC with Primary Sclerosing Cholangitis (PSC) - PSC is a chronic disease characterized by inflammation and scarring of the bile ducts resulting in strictures of the biliary tree; most cases in children are associated with IBD. The diagnosis is made by liver imaging with MRI/MRCP.
* Age <18 years but in adult IBD service
* Intravenous corticosteroids for treatment of colitis within 8 weeks of screening
* Current or previous exposure to tacrolimus, cyclosporin, or mycophenolate,
* Current or previous exposure to biological therapy (anti-TNF, vedolizumab or ustekinumab) and oral JAK-inhibitors (tofacitinib)
* Subjects with current barriers in language or communication that in the judgement of local PI will impede the completion of the trial.
* Female patient with child-bearing potential who does not wish to use a medically acceptable method of contraception throughout the treatment period and for 1 month after discontinuation of treatment. (Appropriate methods of contraception include IUD, oral contraceptive, subdermal implant and double barrier (condom with a contraceptive sponge or contraceptive pessary)
* Pregnancy (current declared or positive urine pregnancy test) or attempting to become pregnant during trial period) or breastfeeding
* A history of overdose, or significant active mental health problems.
* Monogenic IBD (an autosomal condition with an IBD-like phenotype; most common in those with IBD diagnosed <2 years of age)
* Subjects with current - or recent history of - severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, metabolic (including uncontrolled hypercholesterolemia), endocrine, pulmonary, cardiac, neurological disease
* Subjects with a known allergy/contraindication to MitoQ.
* Subjects currently taking any products containing Mitoquinol mesylate (Coenzyme Q10) or any products containing Coenzyme derivatives such as Coenzyme A (CoA, SCoA, CoASH). If subjects are on these products, they can enter the trial after a 7-day washout period.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 24 weeks
  Feasibility of a multi-centre placebo-controlled RCT of an add-on therapy in paediatric UC by the rate of participants recruited per centre over the 15 month recruitment period. Further feasibility parameters such as retention, , adherence and compliance, plus trial and drug acceptability will be assessed. Secondary outcome measures include clinical response and remission at Weeks 6 and 12; and remission, response, reductions in faecal calprotectin and steroid burden, quality of life, safety and tolerance) will be determined at Week 24.

SECONDARY OUTCOMES:
Clincial Response | 6, 12, 24 weeks
  At Weeks 6, 12 and 24 measured using the validated paediatric UC disease activity score 'PUCAI' (drop in PUCAI score >20 points or drop of <20 with absolute score <10 points)
Clinical remission | 6, 12, 24 weeks
  At weeks 6, 12 and 24 (defined as a PUCAI score <10 points.
Clinical response and remission | 6, 12, 24 weeks
  score of 2 or less + no subscore >1) at weeks 6, 12 and 24 on partial Mayo score (9 point score)
Difference in mean PUCAI scores at weeks 6, 12 and 24 weeks | 6, 12, 24 weeks
Steroid-free remission rate at weeks 12 and 24 | 12 and 24 weeks
Steroid-free remission rate at week 24 | 24 weeks
Anti-TNF-free remission rate at week 24 | 24 weeks
Rate of new start iv and/or oral steroid course by week 24 | 24 weeks
Rate of new start immunomodulator (thiopurine/calcineurin inhibitor) by week 24 | 24 weeks
Rate of new start of biological (anti-TNF, vedolizumab, ustekinumab) by week 24 | 24 weeks
Proportions of participants with primary treatment failure with 24 week study period requiring escalation in medical treatment as below: | 24 weeks
  1. (i) Mini-MARVEL M - treatment with oral or intravenous corticosteroids (ii) Mini-MARVEL S - Re-treatment with oral or intravenous corticosteroids
  2. Biologics (anti-TNF, anti-α4β7, anti-IL23 and oral Jak-inhibitors)
  3. Azathioprine or 6-mercaptopurine in participants who were not on a thiopurine at baseline
  4. Oral or intravenous ciclosporin OR oral tacrolimus
Reduction of stool calprotectin of >50% compared to baseline or near normalization (<250ug/g) of faecal calprotectin at week 12 and 24 | 12 and 24 weeks
Mucosal healing with faecal calprotectin <100ug/g at week 12 and at week 24 | 12 and 24 weeks
Cumulative steroid dose baseline to week 24 (steroid burden) | 4 weeks
Quality of life (QoL) - the scores and change from baseline in the validated paediatric IBD quality-of-life score IMPACT 3 at week 12 and week 24 | 12 and 24 weeks
PROM (TUMMY UC) - the scores and change from baseline in the validated TUMMY UC score at week 12 and week 24 | 12 and 24 weeks
Rate and durations of UC-related hospitalizations | 24 weeks
Rate of colectomy for UC or UC-related complications | 24 weeks
Incidence and severity of adverse events/reactions and serious adverse events/reactions | 24 weeks
Drug concentration analyses and research into biomarkers (mitochondrial DNA and formylated peptides) at Baseline, Week 12 and Week 24, plus pharmacogenomics (via DNA sample at Baseline) | 12 and 24 weeks
Precision of the between group effect size (d) - this will be measured by the 95% confidence intervals (CI) around d. | 24 weeks
Achievement of clinically meaningful effect with add-on therapy - we will evaluate if we can gain an estimate of size of clinically meaningful effect between MitoQ and placebo as add-on therapy | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No